CLINICAL TRIAL: NCT00443482
Title: A Randomized, Multi-centre, Double-blind, Double Dummy Placebo Controlled Single-dose Cross-over Study to Demonstrate That 12 and 24 µg of Formoterol Delivered by Concept1 Has a Bronchodilator Efficacy Which is Equivalent to the Same Dose of Formoterol Delivered by Aerolizer in Adult Patients With Persistent Asthma
Brief Title: Study to Demonstrate Equivalence of Formoterol 12 and 24 µg Delivered Via Two Types of Single Dose Dry Powder Inhalers (Concept1 and Aerolizer)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CFOR258D2201
Record Dates: First submitted 2007-03-05; First posted 2007-03-06 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: Asthma; adults; B2 agonist; formoterol
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate

INTERVENTIONS:
Drug: formoterol

SUMMARY:
This study is designed to demonstrate that formoterol 12µg and 24µg delivered by a new inhalation device (Concept1) are equivalent to the corresponding dose of formoterol delivered by the Aerolizer device in terms of efficacy, in patients with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* History of asthma attacks
* Forced expiratory volume in 1 second (measure of how well the lungs are working) is greater than 60% of the predicted value

Exclusion Criteria:

* Asthma is not stable: patients were admitted to hospital or received emergency room treatment
* Patients whose asthma drugs need changing within the month prior to the start of the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
• Efficacy assessed by 12 hour Area Under the Curve (AUC) of FEV1 (forced expiratory volume in 1 second, is a measure of how well the lungs are working)

SECONDARY OUTCOMES:
• Efficacy assessed by forced expiratory volume in 1 second at pre-dose, 15, 30 minutes, 1, 2, 3, 4, 6, 8, 10, 11 and 12 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma AG, Study Director — Novartis Pharmaceuticals
Locations (4):
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bovenden--Lengler
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Wiesbaden